CLINICAL TRIAL: NCT03968471
Title: Chemotherapy-induced Necrosis in Ewing Sarcoma: Which is the Best Scoring Tool
Brief Title: Chemotherapy-induced Necrosis in Ewing Sarcoma
Status: Completed | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Principal Investigator, Alberto Righi, Principal Investigator, Istituto Ortopedico Rizzoli
Other Study IDs: EW-score
Record Dates: First submitted 2019-05-24; First posted 2019-05-30 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Ewing Sarcoma of Bone

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Scoring tool in Chemotherapy-induced necrosis in Ewing sarcoma — The aim of the present study is to evaluate which is the best scoring tool to determine the histological response to chemotherapy in localized Ewing sarcoma of bone.
  The study will exam all the different systems to evaluate the histological necrosis after neo-adjuvant chemotherapy in all patients with localized Ewing sarcomas of bone surgically treated between 1982 and 2012.

SUMMARY:
This is single institution cases series review of histological and clinical data

DETAILED DESCRIPTION:
Investigators will retrieve from the database of the Rizzoli institute all the cases with a histological diagnosis of Ewing sarcoma from 01 Jan 1982 to 31 Dic 2012

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients surgically treated at Rizzoli Institute from 01 Jan 1982 to 31 Dic 2012
2. Patients with diagnosis of Ewing sarcoma of bone who have had neo-adjuvant chemotherapy
3. Diagnosis of Ewing sarcoma localized

Exclusion Criteria:

1. Metastatic disease at presentation
2. Soft tissue origin
3. Radiotherapy before surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Male and female patients surgically treated at Rizzoli Institute from 01 Jan 1982 to 31 Dic 2012 with diagnosis of Ewing sarcoma
Sampling Method: Non-Probability Sample
Enrollment: 474 (Actual)
Dates: Start 2019-05-13 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-01-15 (Actual)

PRIMARY OUTCOMES:
retrospective analysis of cases of Ewing sarcomas | at baseline (Day0)
  Investigators will exam the histological response to chemotherapy in localized Ewing sarcoma of bone and correlate it to clinical outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Righi, MD, Principal Investigator — Istituto Ortopedico Rizzoli IRCCS
Locations (1):
- Dept. of Pathology of IRCCS Istituto Ortopedico Rizzoli, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Esiashvili N, Goodman M, Marcus RB Jr. Changes in incidence and survival of Ewing sarcoma patients over the past 3 decades: Surveillance Epidemiology and End Results data. J Pediatr Hematol Oncol. 2008 Jun;30(6):425-30. doi: 10.1097/MPH.0b013e31816e22f3. PMID 18525458
- [Result] Smith MA, Seibel NL, Altekruse SF, Ries LA, Melbert DL, O'Leary M, Smith FO, Reaman GH. Outcomes for children and adolescents with cancer: challenges for the twenty-first century. J Clin Oncol. 2010 May 20;28(15):2625-34. doi: 10.1200/JCO.2009.27.0421. Epub 2010 Apr 19. PMID 20404250
- [Result] Whelan J, Le Deley MC, Dirksen U, Le Teuff G, Brennan B, Gaspar N, Hawkins DS, Amler S, Bauer S, Bielack S, Blay JY, Burdach S, Castex MP, Dilloo D, Eggert A, Gelderblom H, Gentet JC, Hartmann W, Hassenpflug WA, Hjorth L, Jimenez M, Klingebiel T, Kontny U, Kruseova J, Ladenstein R, Laurence V, Lervat C, Marec-Berard P, Marreaud S, Michon J, Morland B, Paulussen M, Ranft A, Reichardt P, van den Berg H, Wheatley K, Judson I, Lewis I, Craft A, Juergens H, Oberlin O; Euro-E.W.I.N.G.99 and EWING-2008 Investigators. High-Dose Chemotherapy and Blood Autologous Stem-Cell Rescue Compared With Standard Chemotherapy in Localized High-Risk Ewing Sarcoma: Results of Euro-E.W.I.N.G.99 and Ewing-2008. J Clin Oncol. 2018 Sep 6;36(31):JCO2018782516. doi: 10.1200/JCO.2018.78.2516. Online ahead of print. PMID 30188789
- [Result] Picci P, Bohling T, Bacci G, Ferrari S, Sangiorgi L, Mercuri M, Ruggieri P, Manfrini M, Ferraro A, Casadei R, Benassi MS, Mancini AF, Rosito P, Cazzola A, Barbieri E, Tienghi A, Brach del Prever A, Comandone A, Bacchini P, Bertoni F. Chemotherapy-induced tumor necrosis as a prognostic factor in localized Ewing's sarcoma of the extremities. J Clin Oncol. 1997 Apr;15(4):1553-9. doi: 10.1200/JCO.1997.15.4.1553. PMID 9193352
- [Result] Paulussen M, Craft AW, Lewis I, Hackshaw A, Douglas C, Dunst J, Schuck A, Winkelmann W, Kohler G, Poremba C, Zoubek A, Ladenstein R, van den Berg H, Hunold A, Cassoni A, Spooner D, Grimer R, Whelan J, McTiernan A, Jurgens H; European Intergroup Cooperative Ewing's Sarcoma Study-92. Results of the EICESS-92 Study: two randomized trials of Ewing's sarcoma treatment--cyclophosphamide compared with ifosfamide in standard-risk patients and assessment of benefit of etoposide added to standard treatment in high-risk patients. J Clin Oncol. 2008 Sep 20;26(27):4385-93. doi: 10.1200/JCO.2008.16.5720. PMID 18802150

DOCUMENTS (1):
  • Study Protocol (2019-03-08): https://cdn.clinicaltrials.gov/large-docs/71/NCT03968471/Prot_000.pdf